CLINICAL TRIAL: NCT01424462
Title: An Open Label, Randomised Healthy Volunteer Study to Assess the Single Dose Safety and Pharmacokinetics of Three Modified Release Dosage Forms of Firategrast
Brief Title: Healthy Volunteer Pilot Study Using 3 Types of Modified Release Formulations of Firategrast to Investigate How Quickly Absorption From the Digestive System Takes Place.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 114107
Record Dates: First submitted 2011-04-14; First posted 2011-08-29 (Estimated); Last update posted 2017-06-20 (Actual); Status verified 2017-06

CONDITIONS: Multiple Sclerosis, Relapsing-Remitting
Keywords: healthy volunteers; firategrast; Pharmacokinetics; modified release
MeSH Terms: conditions — Multiple Sclerosis, Relapsing-Remitting | interventions — Fumigant 93

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Firategrast XRA (Experimental): Low extended release tablet
  Interventions: Drug: B
- Firategrast XRB (Experimental): Medium extended releast tablet
  Interventions: Drug: C
- Firategrast XRC (Experimental): High extended release tablet
  Interventions: Drug: D
- Firategrast IR (Experimental): Immediate Release reference tablet
  Interventions: Drug: A

INTERVENTIONS:
Drug: A — Single dose treatment IR formulation
  Arms: Firategrast IR
Drug: B — Low Extended release single dose
  Arms: Firategrast XRA
Drug: C — Medium extended release formulation
  Arms: Firategrast XRB
Drug: D — High extended release rate single dose
  Arms: Firategrast XRC

SUMMARY:
This study will investigate how 3 new types of drug formulations are absorbed by the body. This study is termed 'open-label', which means volunteers will be aware of which treatment they are receiving. The study involves all volunteers receiving all 3 different formulations, as a single dose, and there is no placebo (dummy-drug; no active ingredient) in this study. Volunteers will also receive a single dose of a formulation used in previous trials (reference formulation), so as a proper comparison with the new formulations can be made. One of the new formulations will also be administered along with food, to assess if the drug performs or is absorbed differently.

DETAILED DESCRIPTION:
The present study will investigate the tolerability and pharmacokinetics of single oral doses of firategrast administered as the existing immediate release tablet formulation and as three modified release tablet formulations designed to release drug over differing relase rates. The range of release rates is expected to give preliminary information on the performance of a matrix modified release formulation for use in future efficacy studies.

Subjects will receive each formulation in the fasted state in a randomised 4-part single dose crossover fashion. Based on the review of pharmacokinetic data from at least the first two study sessions, subjects may also receive a fifth dose of firategrast, administered after a high fat meal. The formulation administered with food will be chosen based upon pharmacokinetic data from previous dose sessions. Doses administered will be different with respect to gender; the doses are expected to result in similar exposures across the genders.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, aged 18 to 65 yrs inclusive
* Healthy, as determined by study physician
* Capable of giving informed consent

Exclusion Criteria:

* Positive drugs of abuse result
* Positive for HIV or Hepatitis B and/or C viruses
* History of alcohol consumption in excess of average recommended weekly intake (more than 21 units for males, more than 14 units for females)
* Participation in a clinical trial within 90 days of scheduled first dose

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2010-04-19 (Actual); Primary Completion 2010-07-06 (Actual); Study Completion 2010-07-06 (Actual)

PRIMARY OUTCOMES:
Systemic concentration & AUC of study drug | pre-dose, up to 120 hours after each single dose

SECONDARY OUTCOMES:
Adverse events | from screening, through study day, and up to follow-up visit. Spontaneous reporting
Systemic concentration & AUC of study drug metabolite | pre-dose, up to 120 hours after each single dose
Vital signs | screening, pre-dose, up-to 15 hours post does, follow-up visit
12-lead Electrocardiogram | screening, pre-dose and up to 8 hours post dose, then at follow-up
Heamatology, clinical chemistry and Uninalysis | screening, predose, up-to 8 hours post dose, follow-up
  Blood samples for standard clinical safety monitoring, and unine samples

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Randwick, New South Wales, Australia

REFERENCES:
- See also: Results for study 114107 can be found on the GSK Clinical Study Register. — https://gsk-clinicalstudyregister.com/study/114107?search=study&study_ids=114107#rs